CLINICAL TRIAL: NCT06668181
Title: Open-Label, Single-Arm Trial to Evaluate the Pharmacokinetics and Safety of Bimekizumab in Pediatric Study Participants From 2 to Less Than 18 Years of Age With Active Juvenile Idiopathic Arthritis Subtypes Enthesitis-Related Arthritis (Including Juvenile-Onset Ankylosing Spondylitis) and Juvenile Psoriatic Arthritis
Brief Title: An Open-label Study to Evaluate the Pharmacokinetics and Safety of Bimekizumab in Pediatric Study Participants With Active Juvenile Idiopathic Arthritis Subtypes Enthesitis-related Arthritis (Including Juvenile-onset Ankylosing Spondylitis) and Juvenile Psoriatic Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JA0005; U1111-1305-2292 (Other: World Health Organization (WHO)); 2023-508845-41 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Enthesitis-related Arthritis; Juvenile Psoriatic Arthritis
Keywords: Arthritis; Bimekizumab
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bimekizumab (Experimental): Study participants will receive a bimekizumab dose which is dependent on their weight.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Bimekizumab will be administered at pre-specified timepoints.

SUMMARY:
The purpose of this study is to assess plasma bimekizumab concentrations following subcutaneous (sc) bimekizumab administration.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be 2 to <18 years of age inclusive, at the Baseline Visit.
* Study participants who have confirmed diagnosis of enthesitis-related arthritis (ERA; including juvenile-onset ankylosing spondylitis (JAS)) and/or juvenile psoriatic arthritis (JPsA) according to the juvenile-International League of Associations for Rheumatology (JIA-ILAR) classification criteria of at least 3 months duration prior to the Screening Visit.
* Study participants who have active disease (ERA [including JAS] and/or JPsA) defined as having at least 3 active joints, each of which needs to be included in the joints assessed in the JADAS27, and for ERA at least 1 site of enthesitis at Baseline or documented by history.
* Study participants with inadequate response (at least 1 month) or intolerance to at least 1 nonsteroidal anti-inflammatory drug (NSAID).
* Study participants taking concomitant methotrexate or sulfasalazine are allowed to continue the medication if it has been used for the past 12 weeks with a stable dose for the 4 weeks prior to Baseline, with no change in dose for the first 16 weeks of treatment foreseen. (Note: prior or concomitant use of methotrexate or sulfasalazine is NOT required for study participation.)
* Study participants with no concomitant use of second line agents such as disease-modifying and/or immunosuppressive drugs with the exception of methotrexate or sulfasalazine.
* Body weight of ≥10kg.
* Male and female.
* A female study participant will be eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to follow the contraceptive guidance during the Initial Treatment Period, the Open-label Extension (OLE) Period, and for at least 20 weeks after the final dose of investigational medicinal product (IMP; ie, the Safety Follow-up (SFU) Period)
* Capable of giving/having parent(s) or legal representative provide signed informed consent/assent (where appropriate), which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and assent and in this protocol.

Exclusion Criteria:

* Study participants fulfilling any International League of Associations for Rheumatology (ILAR) diagnostic juvenile idiopathic arthritis (JIA) category other than enthesitis-related arthritis (ERA; including juvenile-onset ankylosing spondylitis (JAS)) and/or juvenile psoriatic arthritis (JPsA).
* Study participant has history of inflammatory bowel disease (IBD) or signs/symptoms suggestive of IBD.
* Study participant has active uncontrolled uveitis.
* Study participant has history of active tuberculosis (TB) unless successfully treated, latent TB unless prophylactically treated.
* Study participant has had major surgery (including joint surgery) within the 3 months prior to the Baseline Visit or has planned major surgery within 6 months after entering the study.
* Study participant has laboratory abnormalities at Screening defined in the Protocol.
* Study participant has an active infection or history of infections (such as serious infection, chronic infections, opportunistic infections, unusually severe infections).
* Study participant has received drugs listed in the protocol outside the specified timeframes relative to the Baseline Visit or receives prohibited concomitant treatments.
* Study participant had previous therapy with bimekizumab or prior treatment with other IL-17 biologic response modifier.
* Study participant had prior treatment with more than one biologic response modifier (other than an IL-17).
* Presence of active suicidal ideation, or positive suicide behavior.
* Study participant has been diagnosed with severe depression in the past 6 months.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2028-04-12 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Plasma bimekizumab concentrations over the Initial Treatment Period | Up to Week 16
  Plasma samples will be collected at pre-specified timepoints for measurement of plasma bimekizumab concentrations over the Initial Treatment Period.

SECONDARY OUTCOMES:
Incidence of Treatment-emergent adverse events (TEAEs) | From Baseline (Week 0) to End of Safety Follow-up (up to 141 weeks)
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP.
Incidence of Serious TEAEs | From Baseline (Week 0) to End of Safety Follow-up (up to 141 weeks)
  A SAE is defined as any untoward medical occurrence that, at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent disability/incapacity
  * Is a congenital anomaly/birth defect
  * Important medical events
Incidence of TEAEs leading to discontinuation of investigational medicinal product (IMP) | From Baseline (Week 0) to End of Safety Follow-up (up to 141 weeks)
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP.
Incidence of TEAEs leading to withdrawal from the study | From Baseline (Week 0) to End of Safety Follow-up (up to 141 weeks)
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP.
Incidence of selected safety events of interest (including infection [serious, opportunistic, fungal, and tuberculosis (TB)], inflammatory bowel disease [IBD], and injection site reactions) | From Baseline (Week 0) to End of Safety Follow-up (up to 141 weeks)
  Safety topics of interest are infections (serious, opportunistic, fungal, and tuberculosis), inflammatory bowel disease, and injection site reactions.
Change from Baseline in vital signs (systolic and diastolic blood pressure) at Week 16 | Baseline and Week 16
  Blood pressure will be measured in millimeters of mercury (mmHg).
Change from Baseline in vital signs (heart rate) at Week 16 | Baseline and Week 16
  Heart rate will be measured in beats per minute (beats/min).
Change from Baseline in biochemistry parameters (alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyltransferase) at Week 16 | Baseline and Week 16
  Alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase and gamma-glutamyltransferase will be measured in units per liter (U/L).
Change from Baseline in biochemistry parameters (glucose, potassium, sodium, calcium) at Week 16 | Baseline and Week 16
  Glucose, potassium, sodium and calcium will be measured in millimoles per liter (mmol/L).
Change from Baseline in biochemistry parameters (total bilirubin and direct bilirubin, total protein, blood urea nitrogen, and creatinine) at Week 16 | Baseline and Week 16
  Biochemistry parameters will be measured in micromols per liter (μmol/L).
Change from Baseline in hematology parameters (hemoglobin) at Week 16 | Baseline and Week 16
  Hemoglobin will be measured in grams per liter (g/L).
Change from Baseline in hematology parameters (hematocrit) at Week 16 | Baseline and Week 16
  Hematocrit will be measured in volume percentage (%) of red blood cells in blood.
Change from Baseline in hematology parameters (erythrocytes) at Week 16 | Baseline and Week 16
  Erythrocytes will be measured in number of red blood cells per liter (10^12/L).
Change from Baseline in hematology parameters (platelets, leukocytes neutrophils, lymphocytes, eosinophils, basophils, and monocytes) at Week 16 | Baseline and Week 16
  Platelets, leukocytes, neutrophils, lymphocytes, eosinophils, basophils, and monocytes will be measured in number of white blood cells per liter (10^9/L).
Change from Baseline in growth assessments (height) at Week 16 | Baseline and Week 16
  Growth assessment, as assessed by the change from Baseline in height will be measured in centimeters (cm).
Change from Baseline in growth assessments (weight) at Week 16 | Baseline and Week 16
  Growth assessment, as assessed by the change from Baseline in weight will be measured in kilograms (kg).
Acceptability assessments by injection site pain adverse events (AEs) during the Initial Treatment Period (Week 0 to Week 16) | Week 0 to Week 16
  Incidence rate of injection site pain AEs during the ITP will be reported.
American College of Rheumatology pediatric (ACR Pedi) 30/50/70/90/100 response at Week 16 | Week 16
  ACR assessments are based on a 30%, 50%, 70%, 90%, 100% or greater improvement (for ACR Pedi 30/50/70/90/100 respectively) in at least 3 of the 6 core set measures with no more than 1 of the remaining worsened by >30%. The 6 core set measures are:
  * Number of joints with active arthritis (joints with swelling not due to deformity or inactive synovitis, or joints with limitation of motion with pain, tenderness, or both)
  * Number of joints with limitation of range of motion
  * Physician's Global Assessment of Disease Activity
  * CHAQ total score (Disability Index) completed by parent or caregiver
  * Parent/caregiver global assessment of overall well being of study participant
  * Acute phase reactant (hs-CRP)
Change from Baseline in Juvenile Arthritis Disease Activity Score (JADAS27) -high sensitivity C-reactive protein (hs-CRP) at Week 16 | Baseline and Week 16
  The JADAS27-hs-CRP is a composite disease activity score based on 4 core measures:
  * Number of joints with active arthritis
  * Physician's Global Assessment of Disease Activity
  * Parent/caregiver global assessment of overall well being of study participant
  * Acute phase reactant (hs-CRP); inflammation biomarker. The JADAS27-hs-CRP is calculated as the sum of the scores of the 4 components with a total score range of 0 to 57.
Anti-bimekizumab antibody and neutralizing antibody detection prior to and following IMP administration during the Initial Treatment Period | Up to Week 16
  Anti-bimekizumab antibody and neutralizing antibody detection prior to and following IMP administration during the Initial Treatment Period.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (23):
- Canada (3):
  - Ja0005 50646, Calgary
  - Ja0005 50644, Montreal
  - Ja0005 50645, Saskatoon
- France (4):
  - Ja0005 40777, Indre-et-Loire
  - Ja0005 40510, Le Kremlin-Bicêtre
  - Ja0005 40778, Paris
  - Ja0005 40776, Poitiers
- Germany (7):
  - Ja0005 40369, Berlin
  - Ja0005 40356, Dresden
  - Ja0005 40072, Freiburg im Breisgau
  - Ja0005 40852, Hamburg
  - Ja0005 40787, Sankt Augustin
  - Ja0005 40779, Sendenhorst
  - Ja0005 40427, Tübingen
- Poland (2):
  - Ja0005 40720, Krakow
  - Ja0005 40780, Sosnowiec
- Spain (3):
  - Ja0005 40781, Esplugues de Llobregat
  - Ja0005 40100, Madrid
  - Ja0005 40782, Valencia
- United Kingdom (4):
  - Ja0005 40786, Bristol
  - Ja0005 40783, Manchester
  - Ja0005 40785, Nottingham
  - Ja0005 40784, Stroke-on-trent

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org